CLINICAL TRIAL: NCT07128368
Title: Mechanisms of Resistance Exercise Training for Improved Muscle Insulin Sensitivity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mark Pataky, Associate Consultant I Endocrinology, Diabetes and Metabolism, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-011544; K01DK141911 (NIH)
Record Dates: First submitted 2025-08-13; First posted 2025-08-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Resistance Training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance Exercise Training (Experimental)
  Interventions: Other: Resistance Exercise Training

INTERVENTIONS:
Other: Resistance Exercise Training — Participants will undergo resistance exercise training 3 days a week for approximately 1 hour each day for 8 weeks.

SUMMARY:
To uncover the underlying mechanisms of resistance exercise training benefits on glucose metabolism and insulin sensitivity in muscle.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (≤30min of physical activity on ≤1 day/week)
* Weight stable for ≥3 months prior to study

Exclusion Criteria:

* Active coronary artery disease or heart failure.
* Participation in a structured exercise program > 1 day/week.
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  * Abnormal liver function test results (Transaminase >2 times the upper limit of normal)
  * Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2); If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
  * Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L); testing required within three months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise
  * Abuse of alcohol or recreational drugs
  * Active tobacco usage
  * Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis).
  * Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg) at the time of screening.
  * A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
  * Active pregnancy
  * Menopause (defined as absence of menstruation for 12 consecutive months)
  * Restrictions on Use of Other Drugs or Treatments:

    * Any other medication believed to be a contraindication to the subject's participation.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in muscle protein synthesis | Baseline; 8 weeks
  Rate of insulin-stimulated synthesis of individual proteins

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pataky, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No